CLINICAL TRIAL: NCT03740724
Title: A Phase 1/2 Study of a Combination of FCX-013 (Genetically-Modified Autologous Human Dermal Fibroblasts) Plus Veledimex for the Treatment of Moderate to Severe Localized Scleroderma (Morphea)
Brief Title: A Study of FCX-013 Plus Veledimex for the Treatment of Moderate to Severe Localized Scleroderma (Morphea)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Castle Creek Biosciences, LLC. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FI-SC-001
Record Dates: First submitted 2018-11-06; First posted 2018-11-14 (Actual); Results first posted 2022-06-24 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Morphea; Scleroderma, Localized; Scleroderma
Keywords: Morphea
MeSH Terms: conditions — Scleroderma, Localized; Scleroderma, Diffuse | interventions — veledimex; Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- FCX-013 + veledimex (Experimental): Following the injection of FCX-013, subjects will initiate a 14-day course of veledimex to be taken orally daily
  Interventions: Genetic: FCX-013; Drug: veledimex

INTERVENTIONS:
Genetic: FCX-013 — FCX-013 is a genetically modified cell product obtained from the subject's own skin cells (autologous fibroblasts). The cells are expanded and genetically modified to express metalloproteinase-1 (MMP-1) under the control of a RheoSwitch (RTS®) system. FCX-013 cell suspension is injected intradermally.
  Other Names: Genetically-Modified Autologous Human Dermal Fibroblasts
Drug: veledimex — Veledimex, is a small molecule which activates the RTS to induce expression of MMP-1 and is and provided as a liquid filled gelatin capsule for oral administration
  Other Names: a small-molecule activator ligand for the RheoSwitch (RTS®) system

SUMMARY:
A two-component therapeutic consisting of FCX-013 and veledimex for the treatment of localized scleroderma (or morphea). The first component, FCX-013, is autologous human fibroblasts genetically-modified using lentivirus and encoded for matrix metalloproteinase 1 (MMP-1), a protein responsible for breaking down collagen. FCX-013 is designed to be injected under the skin at the location of the fibrotic lesions where the genetically-modified fibroblast cells will produce MMP-1 to break down excess collagen accumulation. With the FCX-013 therapy, the patient will take an oral compound (Veledimex) to induce MMP-1 protein expression from the injected cells. Once the fibrosis is resolved, the patient will stop taking the oral compound which will stop further MMP-1 production from the injected cells. FCX-013 plus veledimex is being developed in anticipation of improving skin function in patients by resolving fibrotic lesions and normalizing dermal collagen production

DETAILED DESCRIPTION:
Castle Creek is developing a two-component therapeutic product for the treatment of moderate to severe localized scleroderma (morphea). The first component is FCX-013, an autologous genetically modified human dermal fibroblast (GM-HDFs) cell product that is genetically modified with a lentiviral vector (LV) to express human matrix metalloproteinase 1 (MMP1). MMP1 is also known as interstitial collagenase or fibroblast collagenase and is an enzyme that under normal physiological conditions breaks down the extracellular matrix. Specifically, MMP1 breaks down interstitial collagens, types I, II and III. In addition, the FCX-013 cells are also transduced with genetic constructs that encode the RheoSwitch Therapeutic System® (RTS®) an inducible promotor system that in the presence of a small molecule activator ligand controls expression of the MMP1 gene. The RTS® is activated to express MMP1 by the oral administration of the small molecule component. The purpose of this open-label single arm Phase 1/2 study is to investigate the safety and effectiveness of FCX-013 plus veledimex.

ELIGIBILITY:
Inclusion Criteria:

* Subject is an adult, ≥ 18 years of age with moderate to severe localized scleroderma/morphea with sclerotic lesions which have been unresponsive to standard of care therapy.
* Subject has stable control of localized disease (clinically inactive) over the 3 months prior to Screening and through Baseline
* Subject has not participated in previous clinical research study in the 3 months prior to Screening and through Baseline
* Subject has provided informed written consent
* Female subjects of childbearing potential and male subjects engaging in sexual activity that could lead to pregnancy agree to use adequate birth control regimen
* Subject is able to understand the study, cooperate with the study procedures and willing to return to the clinic for the required follow-up visits

Exclusion Criteria:

* Subject has a clinically significant skin disorder other than localized scleroderma/morphea in the anatomical area of interest
* Subject has localized scleroderma/morphea only located on the face or over a joint, or lesions that can be successfully managed with topical medications or phototherapy
* Subject has symptoms consistent with systemic scleroderma that have not been stable, or that require treatment that has not been stable for 3 months prior to Screening and through Baseline
* Subject has been treated with UVA1 phototherapy within 2 months prior to Baseline
* Subject requires treatment with a non-stable regimen of systemic immunosuppressive therapy, for any medical condition, or plans to initiate such treatment during the study period
* Subject requires treatment with a non-stable regimen of physical therapy, for localized scleroderma/morphea, or plans to initiate such treatment during the study period.
* Subject has any medical instability limiting ability to travel to the investigative center.
* Subject has clinical signs of infection at (or in close proximity to) the target lesion.
* Subject has a history of, or current, malignancy at/near site of injection (except basal cell carcinoma or squamous cell carcinoma that have been treated)
* Subject has a history of, or current, clinically significant liver abnormalities.
* Subject has a history of, or current, clinically significant cardiac abnormalities, or a significant abnormality on ECG
* Subject has clinically significant laboratory abnormalities
* Subject has active infection with human immunodeficiency virus (HIV), or hepatitis B/C
* Subject has an active drug or alcohol addiction
* Subject has any known allergy to any of the constituents of the product
* Subject has received an interventional chemical or biological investigational study product for the specific treatment of localized scleroderma in the 3 months prior to Screening and through Baseline
* Subject is pregnant or nursing or plans to become pregnant or nurse during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-12-18 (Actual); Primary Completion 2020-09-23 (Actual); Study Completion 2022-04-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Director, Study Director — Castle Creek Biosciences, LLC.
Locations (1):
- Paddington Testing Co., Inc., Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- FCX-013 + Veledimex: Following the injection of FCX-013, subjects will initiate a 14-day course of veledimex to be taken orally daily
  FCX-013 is a genetically modified cell product obtained from the subject's own skin cells (autologous fibroblasts). The cells are expanded and genetically modified to express metalloproteinase-1 (MMP-1) under the control of a RheoSwitch (RTS®) system. FCX-013 cell suspension is injected intradermally.
  Veledimex, is a small molecule which activates the RTS to induce expression of MMP-1 and is and provided as a liquid filled gelatin capsule for oral administration
Period: Overall Study
Arm/Group | FCX-013 + Veledimex
Started | 1
Completed | 0
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | FCX-013 + Veledimex
Number analyzed (Participants) | 1
Age, Continuous [Mean (Full Range); unit: years] | 46 [46 to 46]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Evaluate the Safety of FCX-013 Plus Veledimex
Description: Safety evaluations include assessment of treatment-emergent adverse events (TEAEs), including serious adverse events (SAEs); change in clinical laboratory values; change in vital signs; change in electrocardiograms (ECGs); and incidence of replication-competent lentivirus (RCL) antibodies.
Time Frame: Study initiation through study completion
Population: 1 subject enrolled but lost to follow up. No outcome data were collected.
Arm/Group | FCX-013 + Veledimex
Number analyzed (Participants) | 0

2. Secondary Outcome: Evaluate the Antifibrotic Effects of FCX-013 Plus Veledimex
Description: Evaluate the antifibrotic effects of FCX-013 plus veledimex
Time Frame: Week 4
Population: 1 subject enrolled but lost to follow up. No outcome data were collected.
Arm/Group | FCX-013 + Veledimex
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time the first subject signed the informed consent form until the final visit/contact with the subject and through study completion/termination (approximately 28 months).
Arm/Group | FCX-013 + Veledimex
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FCX-013 + Veledimex (N=1)
Injection site pain (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol (2020-08-10): https://cdn.clinicaltrials.gov/large-docs/24/NCT03740724/Prot_000.pdf